CLINICAL TRIAL: NCT05031936
Title: Comparison of Intravascular Injection Rates During Cervical and Lumbar Medial Branch Block Using Touhy or Quincke Type Needle
Brief Title: : Intravascular Injection Rates During Cervical Medial Branch Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-07-014
Record Dates: First submitted 2021-08-19; First posted 2021-09-02 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Vascular Complications
Keywords: intravascular injection
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Touhy needle group (Active Comparator): cervical medial branch block using touhy needle
  Interventions: Procedure: cervical spinal injection with 0.2% ropivacaine
- Quincke needle group (Placebo Comparator): cervical medial branch block using quincke needle
  Interventions: Procedure: cervical spinal injection with 0.2% ropivacaine

INTERVENTIONS:
Procedure: cervical spinal injection with 0.2% ropivacaine — spinal injections performed in cervical pillar area to relieve chronic neck pain

SUMMARY:
The purpose of this study is to compare using Toughy needle has an advantage of reducing intravascular injection rates during cervical medial branch block.

DETAILED DESCRIPTION:
In previous reports, the use of Toughy needle was thought to reduce the incidence of intravascular injection as low as 2.9% during lumbar transforaminal injection.

Blunt needles with a pencil point tip, such as Whitacre needles, are not as sharp at their tip as are Quincke needles, which have bevels. Toughy or blunt needles may therefore be less likely to penetrate a vessel during a procedure. Hence, we postulated the incidence of intravenous uptake would be significantly lower using a Toughy needle than using a Quincke needle for lumbar medial branch block. To confirm the intravascular injection rates, we used the real time fluoroscopy after injection of contrast medium.

The goal of this study was to compare the incidence of intravascular injection rate betweeen Toughy and Quincke needles using real time fluoroscopy during cervical medial branch block

ELIGIBILITY:
Inclusion Criteria:

* facet joint arthropathy

Exclusion Criteria:

* allergy to local anesthetics or contrast medium
* pregnancy
* spine deformity
* neurologic abnormality

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
incidence of intravascular injection | 1 minute after finishing cervical medial branch block
  incidence of intravascular injection during cervical medial branch block

SECONDARY OUTCOMES:
time required to complete cervical medial branch block | Baseline, 1 second after the completion of cervical medial branch block
  time required to complete cervical medial branch block
radiation amout to complete cervical medial branch block | Baseline, 1 second after the completion of cervical medial branch block
  radiation amout to complete cervical medial branch block

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, Principal Investigator — Keimyung University
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No